CLINICAL TRIAL: NCT01031381
Title: Phase II Study of RAD001 and Bevacizumab in Recurrent Ovarian, Peritoneal, and Fallopian Tube Cancer An Investigator-initiated, Single-institution Trial at Magee-Womens Hospital
Brief Title: Study of RAD001 and Bevacizumab in Recurrent Ovarian, Peritoneal, and Fallopian Tube Cancer
Acronym: RADBEV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Novartis Pharmaceuticals (Industry); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Robert Edwards, Principal Investigator, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-01-RAD001BEV
Record Dates: First submitted 2009-12-10; First posted 2009-12-14 (Estimated); Results first posted 2016-08-30 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-01

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma
Keywords: Recurrent; ovarian; fallopian tube; primary peritoneal; cancer; Recurrent ovarian, fallopian tube, primary peritoneal cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Recurrence; Neoplasms | interventions — Everolimus; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rad001/Bevacizumab (Other): Patients will receive RAD001 by mouth everyday and Bevacizumab IV every 14 days until clinical progression.
  Interventions: Drug: RAD001; Drug: bevacizumab

INTERVENTIONS:
Drug: RAD001 — RAD001 10mg is taken orally (by mouth) once daily on a continuous basis. RAD001 is provided in tablet form and should be taken with a big glass of water on an empty stomach or after a low-fat meal.
  Other Names: everolimus; derivative of rapamycin
Drug: bevacizumab — bevacizumab will be administered intravenously (IV) once every 14 days.
  Other Names: Avastin

SUMMARY:
This study will investigate the efficacy as well as the safety of RAD001 in combination with bevacizumab for recurrent ovarian, peritoneal, and fallopian tube cancer. RAD001 will be taken orally once daily and bevacizumab will be administered once every 14 days. The study will be conducted over a period of about 3 to 4 years.

DETAILED DESCRIPTION:
In this trial, approximately 50 patients will receive the study drug, RAD001 in combination with bevacizumab (Avastin)chemotherapy. RAD001 will be taken orally once daily and bevacizumab will be administered intravenously once every 14 days. In addition to study treatment, a few blood samples and a sample of the patients tumor from a previous surgery if available will be collected for research.

ELIGIBILITY:
Inclusion Criteria:

* Patients may or may not have measurable disease. Measurable disease is defined according to RECIST criteria. If the patient has had previous radiation to the marker lesion(s), there must be evidence of progression since the radiation was completed.
* Minimum of four weeks since any major surgery, completion of radiation, or completion of all prior systemic anticancer therapy (adequately recovered from the acute toxicities of any prior therapy)
* Fasting serum cholesterol ≤300 mg/dL OR ≤7.75 mmol/L AND fasting triglycerides ≤ 2.5 x ULN.
* Performance status £ 2
* Signed informed consent.

Exclusion Criteria:

* Prior treatment with any investigational drug within the preceding 4 weeks
* Chronic treatment with systemic steroids or another immunosuppressive agent
* Patients should not receive immunization with attenuated live vaccines within one week of study entry or during study period
* Uncontrolled brain or leptomeningeal metastases
* Other malignancies within the past 5 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin.
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation
* Uncontrolled diabetes mellitus
* A known history of HIV seropositivity
* Impairment of gastrointestinal function or gastrointestinal disease
* Patients with an active bleeding diathesis or on oral anti-vitamin K medication (except low dose coumadin)
* Women who are pregnant or breast feeding, or women able to conceive and unwilling to practice an effective method of birth control.
* Patients who have received prior treatment with an mTOR inhibitor (sirolimus, temsirolimus, everolimus).
* Patients with a known hypersensitivity to RAD001 (everolimus), other rapamycins (sirolimus, temsirolimus) or excipients, or bevacizumab
* Patients with serious non-healing wound, ulcer, or bone fracture.
* Patients with known hypersensitivity to Chinese hamster ovary cell products or other recombinant human or humanized antibodies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-09; Primary Completion 2014-01 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Edwards, MD, Principal Investigator — University of Pittsburgh, Magee-Womens Hospital, Gynecologic Oncology Division
Locations (1):
- Magee-Womens Hospital of UPMC, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- RAD001 + Bevacizumab: Patients with recurrent ovarian, peritoneal, and fallopian tube cancer who received RAD001 10 mg/day by mouth and bevacizumab 10 mg/kg intravenously
Period: Overall Study
Arm/Group | RAD001 + Bevacizumab
Started | 59
Completed | 50
Not Completed | 9
Not completed — Physician Decision | 3
Not completed — Withdrawal by Subject | 6

BASELINE CHARACTERISTICS:
Arm/Group | RAD001 + Bevacizumab
Number analyzed (Participants) | 50
Age, Continuous [Median (Full Range); unit: years] | 60.5 [28.0 to 82.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 49
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) at 6-months
Description: The percentage of participants who were alive with the disease (cancer) at 6 months after treatment, but whose disease had not worsened/progressed per Response Evaluation Criteria in Solid Tumors (RECIST v1.1).
Time Frame: Up to 36 months (data collection period for the cohort); Up to 6 months for participant
Population: Patients with recurrent ovarian, peritoneal, and fallopian tube cancer who received RAD001 10 mg/day by mouth and bevacizumab 10 mg/kg intravenously every 14 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | RAD001 + Bevacizumab
Number analyzed (Participants) | 50
percentage of participants | 28 [16.67 to 42.71]

2. Secondary Outcome: Total Number of Participants Experienced a Response (Complete Response+Partial Response+Stable Disease)
Description: The number participants who experienced Complete Response+Partial Response+Stable Disease per Response Evaluation Criteria in Solid Tumors (RECIST v1.1).
Time Frame: Within 4 weeks (28 days) of study treatment initiation (baseline)
Population: Patients with recurrent ovarian, peritoneal, and fallopian tube cancer who received RAD001 10 mg/day by mouth and bevacizumab 10 mg/kg intravenously every 14 days + imaging every 8-12 weeks
Measure: Number; unit: participants
Arm/Group | RAD001 + Bevacizumab
Number analyzed (Participants) | 50
participants | 4

ADVERSE EVENTS:
Arm/Group | RAD001 + Bevacizumab
Serious Adverse Events (participants affected / at risk) | 19/50
Other Adverse Events (participants affected / at risk) | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RAD001 + Bevacizumab (N=50)
Cardiac General - Other (Specify, __) (Cardiac disorders) | 1
Hypertension (Cardiac disorders) | 1
Pericardial effusion (non-malignant) (Cardiac disorders) | 1
Dehydration (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Distension/bloating, abdominal (Gastrointestinal disorders) | 1
Fistula, GI, Colon/cecum/appendix (Gastrointestinal disorders) | 1
Ileus, GI (functional obstruction of bowel, i.e., neuroconstipation) (Gastrointestinal disorders) | 1
Mucositis/stomatitis (clinical exam), Oral cavity (Gastrointestinal disorders) | 2
Obstruction, GI, Ileum (Gastrointestinal disorders) | 1
Obstruction, GI, Small bowel NOS (Gastrointestinal disorders) | 3
Hemorrhage, GU, Bladder (Renal and urinary disorders) | 1
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 1
Infection with unknown ANC, Lung (pneumonia) (Infections and infestations) | 2
Infection with unknown ANC, Urinary tract NOS (Infections and infestations) | 1
Muscle weakness, generalized or specific area (not due to neuropathy), Left-sided (Musculoskeletal and connective tissue disorders) | 1
Neurology - Other (Specify, __) (Nervous system disorders) | 1
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 1
Pain, Abdomen NOS (General disorders) | 2
Pain, Rectum (General disorders) | 1
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other (Specify, __) (Respiratory, thoracic and mediastinal disorders) | 2
Thrombosis/thrombus/embolism (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RAD001 + Bevacizumab (N=50)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 7
Blood/Bone Marrow - Other (Specify, __) (Blood and lymphatic system disorders) | 1
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 2
Lymphopenia (Blood and lymphatic system disorders) | 3
Platelets (Blood and lymphatic system disorders) | 4
Hemoglobin (Blood and lymphatic system disorders) | 9
Supraventricular and nodal arrhythmia, Atrial fibrillation (Cardiac disorders) | 1
Supraventricular and nodal arrhythmia, Sinus bradycardia (Cardiac disorders) | 1
Cardiac Arrhythmia - Other (Specify, __) (Cardiac disorders) | 2
Palpitations (Cardiac disorders) | 2
Supraventricular and nodal arrhythmia, Sinus tachycardia (Cardiac disorders) | 3
Hypertension (Cardiac disorders) | 17
Rigors/chills (General disorders) | 2
Sweating (diaphoresis) (General disorders) | 2
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 3
Insomnia (General disorders) | 3
Constitutional Symptoms - Other (Specify, __) (General disorders) | 5
Weight loss (General disorders) | 8
Fatigue (asthenia, lethargy, malaise) (General disorders) | 30
Nail changes (Skin and subcutaneous tissue disorders) | 1
Rash: dermatitis associated with radiation, Chemoradiation (Skin and subcutaneous tissue disorders) | 1
Rash: erythema multiforme (e.g., Stevens-Johnson syndrome, toxic epidermal necrolysis) (Skin and subcutaneous tissue disorders) | 1
Urticaria (hives, welts, wheals) (Skin and subcutaneous tissue disorders) | 1
Wound complication, non-infectious (Skin and subcutaneous tissue disorders) | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 4
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 5
Dermatology/Skin - Other (Specify, __) (Skin and subcutaneous tissue disorders) | 14
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1
Esophagitis (Gastrointestinal disorders) | 1
Fistula, GI, Colon/cecum/appendix (Gastrointestinal disorders) | 1
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 1
Mucositis/stomatitis (clinical exam), Larynx (Gastrointestinal disorders) | 1
Proctitis (Gastrointestinal disorders) | 1
Ascites (non-malignant) (Gastrointestinal disorders) | 2
Hemorrhoids (Gastrointestinal disorders) | 2
Mucositis/stomatitis (clinical exam), Anus (Gastrointestinal disorders) | 2
Mucositis/stomatitis (clinical exam), Rectum (Gastrointestinal disorders) | 2
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 3
Heartburn/dyspepsia (Gastrointestinal disorders) | 3
Dehydration (Gastrointestinal disorders) | 4
Mucositis/stomatitis (functional/symptomatic), Oral cavity (Gastrointestinal disorders) | 4
Distension/bloating, abdominal (Gastrointestinal disorders) | 6
Gastrointestinal - Other (Specify, __) (Gastrointestinal disorders) | 7
Dental: teeth (Gastrointestinal disorders) | 8
Constipation (Gastrointestinal disorders) | 11
Vomiting (Gastrointestinal disorders) | 13
Anorexia (Gastrointestinal disorders) | 17
Nausea (Gastrointestinal disorders) | 20
Diarrhea (Gastrointestinal disorders) | 22
Mucositis/stomatitis (clinical exam), Oral cavity (Gastrointestinal disorders) | 32
Hematoma (Vascular disorders) | 1
Hemorrhage, GI, Anus (Vascular disorders) | 2
Hemorrhage/Bleeding - Other (Specify, __) (Vascular disorders) | 2
Hemorrhage, pulmonary/upper respiratory, Nose (Vascular disorders) | 8
Infection - Other (Specify, __) (Infections and infestations) | 1
Infection (documented) Urinary tract NOS (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils, Bladder (urinary) (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils, Soft tissue NOS (Infections and infestations) | 1
Infection with normal ANC or Grade 1 or 2 neutrophils, Urinary tract NOS (Infections and infestations) | 1
Infection with unknown ANC, Larynx (Infections and infestations) | 1
Infection with unknown ANC, Oral cavity-gums (gingivitis) (Infections and infestations) | 1
Infection with unknown ANC, Pelvis NOS (Infections and infestations) | 1
Infection with unknown ANC, Bladder (urinary) (Infections and infestations) | 2
Infection with unknown ANC, Bronchus (Infections and infestations) | 2
Infection with unknown ANC, Skin (cellulitis) (Infections and infestations) | 2
Infection with unknown ANC, Upper airway NOS (Infections and infestations) | 2
Infection with unknown ANC, Urinary tract NOS (Infections and infestations) | 5
Edema: head and neck (Blood and lymphatic system disorders) | 1
Lymphatics - Other (Specify, __) (Blood and lymphatic system disorders) | 2
Edema: limb (Blood and lymphatic system disorders) | 7
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 1
Phosphate, serum-low (hypophosphatemia) (Investigations) | 1
Potassium, serum-high (hyperkalemia) (Investigations) | 1
Creatinine (Investigations) | 2
Metabolic/Laboratory - Other (Specify, __) (Investigations) | 2
Albumin, serum-low (hypoalbuminemia) (Investigations) | 3
Magnesium, serum-low (hypomagnesemia) (Investigations) | 3
Potassium, serum-low (hypokalemia) (Investigations) | 4
Cholesterol, serum-high (hypercholesteremia) (Investigations) | 5
Glucose, serum-high (hyperglycemia) (Investigations) | 7
Triglyceride, serum-high (hypertriglyceridemia) (Investigations) | 7
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness, generalized or specific area (not due to neuropathy), Extremity-lower (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness, generalized or specific area (not due to neuropathy), Whole body/generalized (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal/Soft Tissue - Other (Specify, __) (Musculoskeletal and connective tissue disorders) | 7
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 1
Mood alteration, Depression (Nervous system disorders) | 1
Neurology - Other (Specify, __) (Nervous system disorders) | 1
Syncope (fainting) (Nervous system disorders) | 1
Neuropathy: sensory (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 4
Mood alteration, Anxiety (Nervous system disorders) | 6
Ocular/Visual - Other (Specify, __) (Eye disorders) | 1
Pain, Anus (General disorders) | 1
Pain, Dental/teeth/peridontal (General disorders) | 1
Pain, Extremity-limb (General disorders) | 1
Pain, Neuralgia/peripheral nerve (General disorders) | 1
Pain, Pelvis (General disorders) | 1
Pain, Rectum (General disorders) | 1
Pain, Stomach (General disorders) | 1
Pain, Urethra (General disorders) | 1
Pain, Vagina (General disorders) | 1
Pain, Bone (General disorders) | 3
Pain, Joint (General disorders) | 3
Pain, Back (General disorders) | 4
Pain, Throat/pharynx/larynx (General disorders) | 4
Pain, Muscle (General disorders) | 6
Pain, Pain NOS (General disorders) | 6
Pain - Other (Specify, __) (General disorders) | 11
Pain, Head/headache (General disorders) | 14
Pain, Abdomen NOS (General disorders) | 21
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 2
Nasal cavity/paranasal sinus reactions (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary/Upper Respiratory - Other (Specify, __) (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Cystitis (Renal and urinary disorders) | 1
Fistula, GU, Ureter (Renal and urinary disorders) | 1
Obstruction, GU, Ureter (Renal and urinary disorders) | 1
Bladder spasms (Renal and urinary disorders) | 2
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 2
Urinary frequency/urgency (Renal and urinary disorders) | 5
Renal/Genitourinary - Other (Specify, __) (Renal and urinary disorders) | 6
Vaginal discharge (non-infectious) (General disorders) | 2
Vaginal mucositis (General disorders) | 3
Flu-like syndrome (General disorders) | 6
Phlebitis (including superficial thrombosis) (Vascular disorders) | 1
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 1
Vascular - Other (Specify, __) (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes